CLINICAL TRIAL: NCT02401347
Title: A Phase II Clinical Trial of the PARP Inhibitor Talazoparib in BRCA1 and BRCA2 Wild Type Patients With Advanced Triple Negative Breast Cancer and Homologous Recombination Deficiency or Advanced HER2 Negative Breast Cancer or Other Solid Tumors With a Mutation in Homologous Recombination Pathway Genes
Brief Title: Phase II Trial of Talazoparib in BRCA1/2 Wild-type HER2-negative Breast Cancer and Other Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Melinda Telli (Other)
Collaborators: BioMarin Pharmaceutical (Industry); Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Melinda Telli, Assistant Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-31913; NCI-2015-00036 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); BRS0050 (Other: OnCore)
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Results first posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Advanced Breast Cancer; HER2/Neu Negative; Triple-Negative Breast Cancer
Keywords: PALB2 mutation; BRIP1 mutation; BARD1 mutation; Rad51c mutation; PTEN mutation; CHEK2 mutation; ATM mutation; NBN mutation; Rad51d mutation; Rad50 mutation; MRE11 mutation; FANC mutation; HRD assay score; ATR mutation
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A - Triple-negative Breast Cancer (Experimental): Participants with advanced triple-negative breast cancer (TNBC) with homologous recombination deficiency (HRD) based on the Myriad HRD Assay.
  Participants receive talazoparib 1 mg by mouth daily.
  Interventions: Drug: Talazoparib Tosylate
- Cohort B - HER2-negative solid tumor (Experimental): Participants with advanced HER2-negative solid tumor with a deleterious hereditary or cancer somatic mutation in one of the following genes:
  PTEN, PALB2, CHEK2, ATM, NBN, BARD1, BRIP1, RAD50, RAD51C, RAD51D, MRE11, ATR, Fanconi anemia complementation group of genes.
  Participants receive talazoparib 1 mg by mouth daily.
  Interventions: Drug: Talazoparib Tosylate

INTERVENTIONS:
Drug: Talazoparib Tosylate — Participants receive Talazoparib tosylate at 1 mg by mouth daily.
  Other Names: BMN 673

SUMMARY:
The aim of this single-arm phase 2 clinical trial is to evaluate the anti-cancer activity of Talazoparib (also known as BMN 673) in patients with advanced breast cancer with specific genetic or tumor genomic alterations. Patients with either triple-negative or HER2-negative breast cancer are eligible.

DETAILED DESCRIPTION:
Talazoparib (BMN 673) is a novel, dual-mechanism PARP inhibitor that potently inhibits the PARP enzyme and effectively traps PARP on DNA. Talazoparib has shown promising single-agent anti-tumor efficacy in several BRCA1/2 mutation-associated advanced cancers. The efficacy of PARP inhibition in BRCA1/2 wild-type TNBC with homologous recombination (HR) defects and in breast tumors with mutations in other non-BRCA1/2 HR pathway genes is currently unknown.

This phase 2 trial explores the activity of single agent talazoparib in BRCA1/2 wild-type BC patients using an optimal Simon two-stage design. Eligible subjects will be assigned to one of two parallel cohorts: 1) Cohort A: Subjects (n=29) with advanced TNBC with underlying HR defects as assessed by the HRD assay and, 2) Cohort B: Subjects (n=29) with advanced HER2-negative BC with a somatic or germline mutation in a non-BRCA1/2 HR pathway gene. Gene mutations of interest are: PTEN, PALB2, CHEK2, ATM, NBN, BARD1, BRIP1, RAD50, RAD51C, RAD51D, MRE11, ATR, Fanconi anemia complementation group of genes (FANCA, FANCC, FANCD2, FANCE, FANCF, FANCG, FANCL).

ELIGIBILITY:
INCLUSION CRITERIA:

* No deleterious germline BRCA1 or BRCA2 mutation based on full sequencing and comprehensive rearrangement testing at an external reference laboratory; patients with variants of unknown significance will be eligible
* Measurable disease per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1
* Must have progressed on at least 1 prior chemotherapy regimen for the treatment of advanced breast cancer; there is no upper limit on the number of prior therapies
* If prior platinum agent (eg, carboplatin or cisplatin) has been administered, no evidence of progression, or within 8 weeks of stopping platinum treatment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN); if liver function abnormalities are due to hepatic metastasis, then AST and ALT ≤ 5 x ULN
* Total serum bilirubin ≤ 1.5 x ULN (≤ 3 x ULN for Gilbert's syndrome)
* Calculated creatinine clearance ≥ 30 mL/min or serum creatinine ≤ 1.5 mg/dL
* Hemoglobin ≥ 9.0 g/dL with last transfusion at least 14 days before day 1 of study drug
* Absolute neutrophil count (ANC) ≥ 1500/mm^3
* Platelet count ≥ 100,000/mm^3
* Able to take oral medications
* Willing and able to provide written, signed informed consent after the nature of the study has been explained, and prior to any research-related procedures
* Sexually active patients of childbearing potential must be willing to use an acceptable method of contraception such as an intrauterine device or double barrier contraception during treatment and for 30 days after the last dose of study drug
* Females of childbearing potential must have a negative serum pregnancy test at screening and be willing to have additional serum pregnancy tests during the study; females considered not of childbearing potential include those who have been in menopause at least 2 years, or had tubal ligation at least 1 year prior to screening, or who have had total hysterectomy
* Willing and able to comply with all study procedures
* COHORT A SPECIFIC ELIGIBILITY CRITERIA:

  * Histologically-confirmed metastatic or recurrent triple-negative breast cancer (defined as estrogen receptor ≤ 5%, progesterone receptor ≤ 5%, HER2-negative via immunohistochemistry [IHC] or fluorescent in situ hybridization [FISH])
  * An homologous recombination deficiency (HRD) score ≥ 42 on the HRD Assay as assessed on a tumor biopsy sample; in the case that obtaining an adequate metastatic tumor biopsy is not possible, we will assess the HRD score from the primary breast tumor
* COHORT B SPECIFIC ELIGIBILITY CRITERIA:

  * Histologically-confirmed metastatic or recurrent HER2-negative (via IHC or FISH) breast cancer or other histologically-confirmed metastatic solid tumor
  * Deleterious germline or somatic mutation implicated in the homologous recombination (HR) pathway, excluding BRCA1 or BRCA2, based on germline multiplex gene testing or direct tumor next generation DNA sequencing. Genes of interest include: PTEN, PALB2, CHEK2, ATM, NBN, BARD1, BRIP1, RAD50, Rad51c, Rad51d, MRE11, ATR, FANCA, FANCC, FANCD2, FANCE, FANCF, FANCG, FANCL, plus other HR-related genes at the discretion of the primary investigators.

EXCLUSION CRITERIA:

* Any patient with a deleterious mutation in BRCA1 or BRCA2
* Hormone receptor positive and/or HER2 positive breast cancer (Cohort A only)
* HER2 positive breast cancer (Cohort B only)
* Prior treatment with a PARP inhibitor
* Non-measurable disease only
* Pregnant or nursing patients
* Any anti-cancer therapy within the past 21 days of the first day of treatment
* Brain or central nervous system (CNS) metastases

  * Exception: Adequately treated brain metastases documented by baseline computed tomography (CT) or magnetic resonance imaging (MRI) scan that have not progressed since previous scans and do not require corticosteroids (except prednisone ≤ 5 mg/day or equivalent) for management of CNS symptoms. A repeated CT or MRI following the identification of CNS metastases (obtained at least 2 weeks after definitive therapy) must document adequately treated brain metastases
  * Subjects with leptomeningeal carcinomatosis are not permitted
* Other malignancy that is either active or for which patient has received treatment in the last five years excluding non-melanoma skin cancer and carcinoma in situ of the cervix
* Radiation therapy in the last 14 days
* Known to be human immunodeficiency virus positive
* Known active hepatitis C virus
* Known active hepatitis B virus
* Use of any investigational product or investigational medical device within 28 days before day 1 of study drug
* Major surgery requiring a prolonged hospitalization or recovery within 21 days before day 1 of study drug
* Concurrent disease or condition that would interfere with study participation or safety, such as any of the following:

  * Active, clinically significant infection either grade > 2 by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 or requiring the use of parenteral anti-microbial agents within 7 days before day 1 of study drug
  * Clinically significant bleeding diathesis or coagulopathy, including known platelet function disorders
  * Known hypersensitivity to any of the components of BMN 673

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2022-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melinda L Telli, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Medicine at Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gruber JJ, Afghahi A, Timms K, DeWees A, Gross W, Aushev VN, Wu HT, Balcioglu M, Sethi H, Scott D, Foran J, McMillan A, Ford JM, Telli ML. A phase II study of talazoparib monotherapy in patients with wild-type BRCA1 and BRCA2 with a mutation in other homologous recombination genes. Nat Cancer. 2022 Oct;3(10):1181-1191. doi: 10.1038/s43018-022-00439-1. Epub 2022 Oct 17. PMID 36253484

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A - Triple-negative Breast Cancer: Participants with advanced triple-negative breast cancer (TNBC) with homologous recombination deficiency (HRD) based on the Myriad HRD Assay.
  Participants receive talazoparib 1 mg by mouth daily.
  Talazoparib Tosylate: Participants receive Talazoparib tosylate at 1 mg by mouth daily.
- Cohort B - HER2-negative Solid Tumor: Participants with advanced HER2-negative solid tumor with a deleterious hereditary or cancer somatic mutation in one of the following genes:
  PTEN, PALB2, CHEK2, ATM, NBN, BARD1, BRIP1, RAD50, RAD51C, RAD51D, MRE11, ATR, Fanconi anemia complementation group of genes.
  Participants receive talazoparib 1 mg by mouth daily.
  Talazoparib Tosylate: Participants receive Talazoparib tosylate at 1 mg by mouth daily.
Period: Overall Study
Arm/Group | Cohort A - Triple-negative Breast Cancer | Cohort B - HER2-negative Solid Tumor
Started | 1 | 20
Completed | 1 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A - Triple-negative Breast Cancer | Cohort B - HER2-negative Solid Tumor | Total
Number analyzed (Participants) | 1 | 20 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 15 | 16
  >=65 years | 0 | 5 | 5
Age, Continuous [Median (Standard Deviation); unit: years] | 42.5 (NA) — Cannot compute standard deviation on a single value. | 53.8 (9.6) | 53.6 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 15 | 16
  Male | 0 | 5 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 1 | 19 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 0 | 15 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 20 | 21

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (OR)
Description: Objective response (OR) is a common measure of benefit. OR is defined as the number of participants who achieved complete response (CR) or partial clinical (PR), per the Response Evaluation Criteria in Solid Tumors (RECIST) Criteria (v1.1). RECIST Criteria are assessed by physical measurement; magnetic resonance imaging (MRI); computed tomography (CT), positron emission tomography (PET)-CT; and/or X-rays, as follows:
  * CR = Disappearance of all target and non-target lesions
  * PR = ≥30% decrease in the sum of the long diameter of target lesions
  * OR = CR+PR
  * Stable disease (SD) = Small changes that do not meet any of the above criteria
  * Progressive disease (PD) = ≥20% increase in long diameter of target lesions, and/or the appearance of any new lesion(s) The outcome is expressed as the number of participants that achieved either CR or PR within 24 weeks of the start of treatment, a number without dispersion.
Time Frame: up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A - Triple-negative Breast Cancer | Cohort B - HER2-negative Solid Tumor
Number analyzed (Participants) | 1 | 20
Participants
  Complete response (cR) | 0 | 0
  Partial response (PR) | 0 | 3
  Overall response (CR+PR) | 0 | 3
  Stable disease (SD) | 0 | 7
  Progressive disease (PD) | 1 | 10

2. Secondary Outcome: Clinical Benefit (CB)
Description: Clinical benefit (CB) is a common measure of benefit. CB is defined as the number of participants who achieved complete response (CR); partial clinical (PR); or stable disease (SD), per the Response Evaluation Criteria in Solid Tumors (RECIST) Criteria (v1.1). RECIST Criteria are assessed by physical measurement; magnetic resonance imaging (MRI); computed tomography (CT), positron emission tomography (PET)-CT; and/or X-rays, as follows:
  * CR = Disappearance of all target and non-target lesions
  * PR = ≥30% decrease in the sum of the long diameter of target lesions
  * SD = Small changes that do not meet any of the above criteria
  * CB = CR+PR+SD
  * Progressive disease (PD) = ≥20% increase in long diameter of target lesions, and/or the appearance of any new lesion(s) The outcome is expressed as the number of participants that achieved either CR, PR, or SD within 24 weeks of the start of treatment, a number without dispersion.
Time Frame: up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A - Triple-negative Breast Cancer | Cohort B - HER2-negative Solid Tumor
Number analyzed (Participants) | 1 | 20
Participants
  Complete response (CR) | 0 | 0
  Partial response (PR) | 0 | 3
  Stable disease (SD) | 0 | 7
  Clinical benefit (CB) | 0 | 10
  Progressive disease (PD) | 1 | 10

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) is a common measure of benefit. PFS means to remain alive with disease or tumor progression. Progression was defined per the Response Evaluation Criteria in Solid Tumors (RECIST) Criteria (v1.1) as any ≥20% increase in long diameter of the target lesions, and/or the appearance of any new lesion(s). PFS is expressed as the number of participants who remained alive without progression after 1 year, a number without dispersion.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A - Triple-negative Breast Cancer | Cohort B - HER2-negative Solid Tumor
Number analyzed (Participants) | 1 | 20
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse through 30 days after the last dose of study medication, which had an average duration of 3 cycles (28 days per cycle) and were followed for survival through 1 year.
Arm/Group | Cohort A - Triple-negative Breast Cancer | Cohort B - HER2-negative Solid Tumor
All-Cause Mortality (participants affected / at risk) | 1/1 | 9/20
Serious Adverse Events (participants affected / at risk) | 0/1 | 3/20
Other Adverse Events (participants affected / at risk) | 1/1 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A - Triple-negative Breast Cancer (N=1) | Cohort B - HER2-negative Solid Tumor (N=20)
Thrombocytopenia (Investigations) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Weakness in extremity, right leg, progressing (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Weakness in extremities, right side (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intracranial masses, supratentorial and infratentoria (Nervous system disorders) | 0 (0) | 1 (1)
Pneumothorax, post-lung biopsy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A - Triple-negative Breast Cancer (N=1) | Cohort B - HER2-negative Solid Tumor (N=20)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 4 (4)
Lymphedema (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Deep venous thrombosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 9 (9)
Constipation (Gastrointestinal disorders) | 0 (0) | 7 (7)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 9 (9)
Pain (General disorders) | 0 (0) | 3 (3)
Edema limbs (peripheral edema) (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 2 (2)
Flu-like symptoms (General disorders) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 7 (7)
Alkaline phosphatase increased (Investigations) | 0 (0) | 5 (5)
Neutropenia (Investigations) | 0 (0) | 5 (5)
Thrombocytopenia (Investigations) | 0 (0) | 3 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (3)
Aspartate Amino Transferase increased (Investigations) | 0 (0) | 3 (3)
Weight loss (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Rash, maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/47/NCT02401347/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT02401347/ICF_001.pdf